CLINICAL TRIAL: NCT03509350
Title: A Multi-center, Randomized, Placebo-controlled, Double-blind, Adaptive Clinical Trial of Vitamin C, Thiamine and Steroids as Combination Therapy in Patients With Sepsis.
Brief Title: Vitamin C, Thiamine, and Steroids in Sepsis
Acronym: VICTAS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: The Marcus Foundation (Other)
Responsible Party: Principal Investigator, Jonathan Sevransky, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB00102528; IRB00164053 (Other: Johns Hopkins IRB)
Record Dates: First submitted 2018-04-10; First posted 2018-04-26 (Actual); Results first posted 2020-09-18 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-03

CONDITIONS: Sepsis
Keywords: Vitamin C; Thiamine; Corticosteroid
MeSH Terms: conditions — Sepsis | interventions — Ascorbic Acid; Thiamine; thiamine hydrochloride; Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Protocol (Experimental): Participants randomized to the treatment protocol will receive the VICTAS Intervention, consisting of intravenous vitamin C, thiamine, and hydrocortisone for four days or until ICU discharge.
  Interventions: Drug: Vitamin C; Drug: Thiamine; Drug: Hydrocortisone
- Control Protocol (Placebo Comparator): A placebo to match the VICTAS intervention will be administered for four days or until ICU discharge. During the treatment period, if an indication for steroids exist, the treating physicians are permitted to initiate open-label corticosteroid therapy based on local practice and international guidelines. If this occurs, the hydrocortisone/placebo will be withheld and subjects will be started on open-label corticosteroids.
  Interventions: Drug: Vitamin C Placebo; Drug: Thiamine Placebo; Drug: Hydrocortisone Placebo

INTERVENTIONS:
Drug: Vitamin C — Intravenous vitamin C (1.5 grams every 6 hours) will be administered for 4 days or until ICU discharge.
  Other Names: Ascorbic acid
  Arms: Treatment Protocol
Drug: Thiamine — Intravenous thiamine (100 mg every 6 hours) will be administered for 4 days or until ICU discharge.
  Other Names: Thiamine hydrochloride
  Arms: Treatment Protocol
Drug: Hydrocortisone — Intravenous hydrocortisone (50 mg every 6 hours) will be administered for 4 days or until ICU discharge.
  Other Names: Hydrocortisone sodium succinate
  Arms: Treatment Protocol
Drug: Vitamin C Placebo — A placebo to match intravenous vitamin C (1.5 grams every 6 hours) will be administered for 4 days or until ICU discharge.
  Other Names: Placebo
  Arms: Control Protocol
Drug: Thiamine Placebo — A placebo to match intravenous thiamine (100 mg every 6 hours) will be administered for 4 days or until ICU discharge.
  Other Names: Placebo
  Arms: Control Protocol
Drug: Hydrocortisone Placebo — A placebo to match intravenous hydrocortisone (50 mg every 6 hours) will be administered for 4 days or until ICU discharge. Steroids will be used when clinically indicated.
  Other Names: Placebo
  Arms: Control Protocol

SUMMARY:
The VItamin C, Thiamine And Steroids in Sepsis (VICTAS) Study is a double-blind, placebo-controlled, adaptive randomized clinical trial designed to investigate the efficacy of the combined use of vitamin C, thiamine and corticosteroids versus indistinguishable placebos for patients with sepsis. The objective of this study is to demonstrate the efficacy of combination therapy using vitamin C, thiamine and corticosteroids in reducing mortality and improving organ function in critically ill patients with sepsis.

DETAILED DESCRIPTION:
Sepsis is an inflammatory syndrome with life threatening organ dysfunction resulting from a dysregulated host response to infection. The global burden is estimated to exceed 15 million cases annually. In the United States, the incidence is increasing and currently there are more 1,750,000 cases each year, with more than half requiring intensive care unit (ICU) admission. Further, sepsis cases account for 30%- 50% of all hospital deaths, making it the 3rd leading cause of death in the United States, and is the most expensive reason for hospitalization with annual expenditures exceeding $20 billion. Notably, even among those that do survive, many endure significant reductions in physical, emotional and cognitive quality of life. New therapeutic approaches to reduce the high morbidity and mortality of sepsis are needed.

Current management strategies focus on early aggressive fluid resuscitation, blood pressure support with vasopressors, early appropriate antibiotics, and the identification and control of infected sites. Though outcomes have improved with the bundled deployment of these strategies, mortality remains high at 20 - 30%. Despite over a hundred phase 2 and phase 3 clinical trials of pharmacological agents with the potential to improve sepsis outcomes, only antibiotics have demonstrated reproducible benefits.

The purpose of the current study is therefore to determine (or confirm) the efficacy of the combination therapy consisting of vitamin C, thiamine, and corticosteroids in the management of patients with circulatory and/or respiratory dysfunction resulting from sepsis. This subset of sepsis patients has been chosen because they are easily identified, have a high mortality, and consume significant critical care resources. As such, any improvements in outcomes attributed to effective therapies would be of great value to patients, as well as their care providers and healthcare systems. Further, because the promulgated therapies are composed of three inexpensive and readily available drugs, its efficacy would have important implications the management of sepsis in both well and poorly resourced settings worldwide.

The VItamin C, Thiamine And Steroids in Sepsis (VICTAS) Study is a double-blind, placebo-controlled, adaptive randomized clinical trial designed to investigate the efficacy of the combined use of vitamin C, thiamine and corticosteroids (the Treatment Protocol) versus indistinguishable placebos (the Control Protocol) for patients with sepsis. The trial will enroll up to 2000 participant and employs a novel endpoint that approximates a patient's risk of death based on the time spent on vasopressors or receiving respiratory support. Time spent on vasopressors or receiving respiratory support captures a patient's speed of recovery. Mortality rate is a key secondary endpoint for the trial.

Specific Aims

1. To demonstrate the efficacy of combination therapy using vitamin C, thiamine and corticosteroids to reduce the duration of cardiovascular and respiratory organ dysfunction in critically ill patients with sepsis.
2. To demonstrate the efficacy of combination therapy using vitamin C, thiamine and corticosteroids to reduce 30-day mortality in critically ill patients with sepsis.

Explicit subject consent for participation in long term telephone follow-up will be sought for all patients at all sites. Participation in long term outcome assessments is not required for participation in other aspects of the VICTAS study, i.e., patients may individually opt out of this portion of the study. In these participants a diverse array of neurocognitive outcomes will be assessed approximately 6 months after patient discharge. Evaluations will be done using a specially-designed battery of tests that evaluates key aspects of functioning and behavior and will be administered via phone by the Vanderbilt Long-Term Outcomes team, which will serve as the coordinating center for these follow-up assessments. The battery, which takes about 40 minutes to complete, will assess cognition, mental health, quality of life, and employment - all of which have been shown to be adversely affected in between one third and two thirds of survivors of sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or confirmed infection as evidenced by ordering of blood cultures and administration of at least one antimicrobial agent
* Anticipated or confirmed intensive care unit (ICU) admission
* Acute respiratory or cardiovascular organ dysfunction attributed to sepsis as evidenced by at least one of the following requirements:

  1. Vasopressor Requirement - Continuous infusion of norepinephrine, epinephrine, vasopressin, dopamine, phenylephrine or other vasopressor agents at any dose for greater than 1 hour and required to maintain a mean arterial pressure ≥ 65 mm Hg despite intravenous crystalloid infusion of at least 1000cc
  2. Respiratory Support Requirement - Acute hypoxemic respiratory failure defined as persistent hypoxemia (partial pressure of arterial oxygen (PaO2)/fraction of inspired oxygen (FiO2) ≤ 300 or blood oxygen saturation (SpO2)/FiO2 ≤ 315) requiring (1) intubation and mechanical ventilation, or (2) positive pressure ventilation via tight-fitting face mask (i.e. continuous positive airway pressure (CPAP) or bilevel positive airway pressure (BiPAP) or (3) high flow nasal cannula ≥ 40 liter per minute (LPM) flow and FiO2 ≥ 0.40

Exclusion Criteria:

* Weight < 40 kilograms (kg)
* Prior enrollment in this study
* Qualifying organ dysfunction no longer present at the time subject would be randomized
* Cardiovascular or respiratory organ failure caused by an illness other than sepsis
* First episode of qualifying organ dysfunction during the current emergency department (ED) or ICU admission occurred > 24 hours before the subject could be randomized
* Limitations of care (defined as refusal of cardiovascular and respiratory support modes) including "do not intubate" (DNI) status
* Current hospitalization > 30 days at time of randomization
* Chronic hypoxemia requiring supplemental non-invasive oxygen (nasal cannula or NIPPV) or home mechanical ventilation
* Chronic cardiovascular failure requiring home mechanical hemodynamic support (e.g., LVAD) or home chemical hemodynamic support (e.g., milrinone)
* Known allergy or contraindication to vitamin C, thiamine, and/or corticosteroids (including previously or currently diagnosed primary hyperoxaluria and/or oxalate nephropathy, or known/suspected ethylene glycol ingestion, or known glucose-6-phosphate dehydrogenase (G6PD) deficiency)
* Use of vitamin C at a dose of > 1 gram daily within the 24 hours preceding first episode of qualifying organ dysfunction during a given ED or ICU admission
* Chronic disease/illness that, in the opinion of the site investigator, have an expected lifespan of < 30 days unrelated to current sepsis diagnosis (e.g., stage IV malignancy, neurodegenerative disease, etc.)
* Pregnancy or known active breastfeeding
* Prisoner or Incarceration
* Current participation in another interventional research study
* Inability or unwillingness of subject or legal surrogate/representative to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2020-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Sevransky, MD, MHS, Principal Investigator — Emory University
Locations (43):
- United States (43):
  - Maricopa Integrated Health System, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Stanford University, Stanford, California
  - University of Colorado Denver, Denver, Colorado
  - Denver Health, Denver, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Christiana Care, Newark, Delaware
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - University of Florida Jacksonville, Jacksonville, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Lousiana State University, New Orleans, Louisiana
  - Johns Hopkins Bayview, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Baystate Health, Springfield, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center Weiler, The Bronx, New York
  - Montefiore Medical Center Moses, The Bronx, New York
  - Duke University, Durham, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - University of Cincinnati Physicians Company, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - University of Pennsylvania Health System Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Intermountain Medical Center, Murray, Utah
  - University of Utah, Salt Lake City, Utah
  - Sentara Healthcare, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Bon Secours, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Williams Roberson S, Nwosu S, Collar EM, Kiehl AL, Harrison FE, Bastarache J, Wilson JE, Mart MF, Sevransky JE, Ely EW, Lindsell CJ, Jackson JC; VICTAS Investigators. Association of Vitamin C, Thiamine, and Hydrocortisone Infusion With Long-term Cognitive, Psychological, and Functional Outcomes in Sepsis Survivors: A Secondary Analysis of the Vitamin C, Thiamine, and Steroids in Sepsis Randomized Clinical Trial. JAMA Netw Open. 2023 Feb 1;6(2):e230380. doi: 10.1001/jamanetworkopen.2023.0380. PMID 36853612
- [Derived] Sevransky JE, Rothman RE, Hager DN, Bernard GR, Brown SM, Buchman TG, Busse LW, Coopersmith CM, DeWilde C, Ely EW, Eyzaguirre LM, Fowler AA, Gaieski DF, Gong MN, Hall A, Hinson JS, Hooper MH, Kelen GD, Khan A, Levine MA, Lewis RJ, Lindsell CJ, Marlin JS, McGlothlin A, Moore BL, Nugent KL, Nwosu S, Polito CC, Rice TW, Ricketts EP, Rudolph CC, Sanfilippo F, Viele K, Martin GS, Wright DW; VICTAS Investigators. Effect of Vitamin C, Thiamine, and Hydrocortisone on Ventilator- and Vasopressor-Free Days in Patients With Sepsis: The VICTAS Randomized Clinical Trial. JAMA. 2021 Feb 23;325(8):742-750. doi: 10.1001/jama.2020.24505. PMID 33620405
- [Derived] Lindsell CJ, McGlothlin A, Nwosu S, Rice TW, Hall A, Bernard GR, Busse LW, Ely EW, Fowler AA, Gaieski DF, Hinson JS, Hooper MH, Jackson JC, Kelen GD, Levine M, Martin GS, Rothman RE, Sevransky JE, Viele K, Wright DW, Hager DN. In response: Letter on update to the Vitamin C, Thiamine and Steroids in Sepsis (VICTAS) protocol. Trials. 2020 Apr 22;21(1):351. doi: 10.1186/s13063-020-04290-6. PMID 32317004
- [Derived] Morgan J. Surviving sepsis and intensive care unit delirium: a remarkable recovery. Lancet Respir Med. 2020 Mar;8(3):241-242. doi: 10.1016/S2213-2600(20)30043-6. Epub 2020 Jan 30. No abstract available. PMID 32007132
- [Derived] Lindsell CJ, McGlothlin A, Nwosu S, Rice TW, Hall A, Bernard GR, Busse LW, Ely EW, Fowler AA, Gaieski DF, Hinson JS, Hooper MH, Jackson JC, Kelen GD, Levine M, Martin GS, Rothman RE, Sevransky JE, Viele K, Wright DW, Hager DN. Update to the Vitamin C, Thiamine and Steroids in Sepsis (VICTAS) protocol: statistical analysis plan for a prospective, multicenter, double-blind, adaptive sample size, randomized, placebo-controlled, clinical trial. Trials. 2019 Dec 4;20(1):670. doi: 10.1186/s13063-019-3775-8. PMID 31801567
- [Derived] Hager DN, Hooper MH, Bernard GR, Busse LW, Ely EW, Fowler AA, Gaieski DF, Hall A, Hinson JS, Jackson JC, Kelen GD, Levine M, Lindsell CJ, Malone RE, McGlothlin A, Rothman RE, Viele K, Wright DW, Sevransky JE, Martin GS. The Vitamin C, Thiamine and Steroids in Sepsis (VICTAS) Protocol: a prospective, multi-center, double-blind, adaptive sample size, randomized, placebo-controlled, clinical trial. Trials. 2019 Apr 5;20(1):197. doi: 10.1186/s13063-019-3254-2. PMID 30953543

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant enrollment began on August 22, 2018. Follow-up for the primary outcome measure was completed on August 22, 2019 and follow up for the secondary outcome measures was completed on January 29, 2020. Participants were recruited from multiple sites in the United States of America.
Groups:
- Treatment Protocol: Participants randomized to the treatment protocol received the VICTAS Intervention, consisting of intravenous vitamin C, thiamine, and hydrocortisone for four days or until ICU discharge.
- Control Protocol: Participants in the control group received a placebo to match the VICTAS intervention, which was administered for four days or until ICU discharge.
Period: Overall Study
Arm/Group | Treatment Protocol | Control Protocol
Started | 252 | 249
Completed | 252 | 247
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Protocol | Control Protocol | Total
Number analyzed (Participants) | 252 | 249 | 501
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 148 | 143 | 291
  >=65 years | 104 | 106 | 210
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62 [51 to 69] | 61 [50 to 72] | 62 [50 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 115 | 228
  Male | 139 | 134 | 273
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 24 | 56
  Not Hispanic or Latino | 211 | 215 | 426
  Unknown or Not Reported | 9 | 10 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 70 | 80 | 150
  White | 149 | 135 | 284
  More than one race | 33 | 34 | 67
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 252 | 249 | 501

OUTCOME MEASURES:

1. Primary Outcome: Vasopressor and Ventilator-free Days (VVFD)
Description: The primary outcome measure is VVFD in the first 30 days after the start of treatment. The endpoint was recorded to the nearest day. Participants who died are scored zero days, even if there was a period during which the participant was alive and free of vasopressors and mechanical ventilation. Participants who must return to ventilation and/or vasopressors had their counters reset at zero days.
Time Frame: Up to Day 30
Population: This analysis uses an intent-to-treat (ITT) analysis set, which includes all participants who enrolled in the study.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Treatment Protocol | Control Protocol
Number analyzed (Participants) | 252 | 249
days | 25 [0 to 29] | 26 [0 to 28]

2. Secondary Outcome: Mortality at 30 Days
Description: The number of participants who did not survive until Day 30 is compared between study arms.
Time Frame: Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Protocol | Control Protocol
Number analyzed (Participants) | 252 | 249
Participants | 56 | 60

3. Secondary Outcome: Intensive Care Unit (ICU) Mortality
Description: The number of participants who died while in the ICU is compared between study arms.
Time Frame: Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Protocol | Control Protocol
Number analyzed (Participants) | 252 | 249
Participants | 52 | 49

4. Secondary Outcome: Mortality at 180 Days
Description: The number of participants who did not survive until Day 180 is compared between study arms.
Time Frame: Day 180
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Protocol | Control Protocol
Number analyzed (Participants) | 252 | 249
Participants | 102 | 94

5. Secondary Outcome: Length of ICU Stay
Description: The number of days that participants were in the ICU is compared between study arms.
Time Frame: Day 30
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treatment Protocol | Control Protocol
Number analyzed (Participants) | 252 | 249
days | 6.7 (7.3) | 6.4 (6.9)

6. Secondary Outcome: Length of Hospital Stay
Description: The number of days that participants were in the hospital is compared between study arms.
Time Frame: Day 30
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treatment Protocol | Control Protocol
Number analyzed (Participants) | 252 | 249
days | 12.6 (10) | 13.5 (25.7)

7. Secondary Outcome: Digit Span Test Score
Description: The Digit Span Test is used to assesses attention. In the Digit Span Test, participants are read a series of numbers and are asked to repeat them back in the same order. The Digit Span test is scored by the number of digits the participant is able to remember in each test. Higher scores indicate greater ability to pay attention and to remember sequences. The average adult can remember about 7 numbers, plus or minus two, without making an error.
Time Frame: Day 180
Measure: Mean (Standard Deviation); unit: numbers recalled
Arm/Group | Treatment Protocol | Control Protocol
Number analyzed (Participants) | 252 | 249
numbers recalled | 8.3 (3.1) | 9.5 (3.8)

8. Secondary Outcome: Number of Participants With Delirium Assessed With the DeliriumTelephone Confusion Assessment Method (CAM)
Description: The Telephone CAM evaluates dementia with 9-items, where additional questions are asked if symptoms are present. Rather than providing a summary score, if participants exhibit signs of a change in mental status which fluctuates and they experience inattention, along with disorganized thinking or altered level of consciousness, delirium is suggested.
Time Frame: Day 180
Population: Telephone data are available only on 168 participants
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Protocol | Control Protocol
Number analyzed (Participants) | 86 | 82
Participants | 0 | 0

9. Secondary Outcome: Hayling Test Score
Description: Executive function is assessed with the Hayling Test. The Hayling Test includes two parts of 15 items each where participants complete sentences by providing the missing word. The test is scored as the amount of time it takes, in seconds, to recite a correct response and the appropriateness of the response (in Part 2). Scaled scores range from 1 to 10 where 1 = impaired, 6 = average, and 10 = very superior.
Time Frame: Day 180
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Protocol | Control Protocol
Number analyzed (Participants) | 252 | 249
units on a scale | 4.2 (1.9) | 4.2 (1.8)

10. Secondary Outcome: Controlled Oral Word Association Test (COWAT) Score
Description: Language is assessed with the Controlled Oral Word Association Test (COWAT). Participants generate words beginning with selected letters within 60 seconds. Generating a higher number of words indicates greater language skills.
Time Frame: Day 180
Measure: Mean (Standard Deviation); unit: words
Arm/Group | Treatment Protocol | Control Protocol
Number analyzed (Participants) | 252 | 249
words | 40 (11) | 40 (11)

11. Secondary Outcome: Wechsler Memory Scale III - Delayed Recall Logical Memory Score
Description: Memory is assessed with the Logical Memory subtest from the Wechsler Memory Scale III. Participants listened to two short paragraphs and were asked to recall details from each story after 30 minutes. Scores represent the number of correctly remembered details. Total scores range from 0 to 25 with higher scores reflecting better memory.
Time Frame: Day 180
Measure: Mean (Standard Deviation); unit: correct story details
Arm/Group | Treatment Protocol | Control Protocol
Number analyzed (Participants) | 252 | 249
correct story details | 6.9 (2.8) | 8.1 (3.2)

12. Secondary Outcome: Telephone Interview for Cognitive Status (TICS)
Description: The Telephone Interview for Cognitive Status (TICS) is an 11-item instrument assessing orientation. Correct responses to the items are scored in a variety of ways, depending on how much of the response is correct. Total scores range from 0 to 41 with higher scores indicating increased cognitive orientation.
Time Frame: Day 180
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Protocol | Control Protocol
Number analyzed (Participants) | 252 | 249
score on a scale | 30.6 (4.9) | 31.2 (5.2)

13. Secondary Outcome: Wechsler Adult Intelligence Scale (WAIS)-IV Similarities Score
Description: Reasoning is assessed with the WAIS-IV Similarities instrument. Participants were asked to explain how two words are alike. Responses are scored according to how correct they are, with a score of 0 for incorrect answers. After 3 consecutive scores of 0 the survey is stopped. Total raw scores vary depending on the number of word pairs presented. Higher scores indicate better performance. Scores will be compared between study arms.
Time Frame: Day 180
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Protocol | Control Protocol
Number analyzed (Participants) | 252 | 249
score on a scale | 7.7 (3.3) | 8.2 (3.2)

14. Secondary Outcome: Katz Index of Independence in Activities of Daily Living (ADL) Score
Description: Activities of daily living is assessed with the Katz ADL instrument. The Katz ADL has 6 items asking if participants can perform daily tasks independently. Responses are scored as 1 = yes and 0 = no. Total scores range from 0 to 6 with higher scores indicating greater independence.
Time Frame: Day 180
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Protocol | Control Protocol
Number analyzed (Participants) | 252 | 249
score on a scale | 2.8 (3.9) | 2.4 (3.6)

15. Secondary Outcome: Number of Participants Employed
Description: The Employment Questionnaire is a brief measure of the participant's employment history and ability or capacity to work. The number of participants who indicated being employed are presented here.
Time Frame: Day 180
Population: This analysis includes participants who completed the Employment Questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Protocol | Control Protocol
Number analyzed (Participants) | 99 | 96
Participants | 17 | 25

16. Secondary Outcome: Functional Activities Questionnaire (FAQ) Score
Description: Instrumental activities of daily living is assessed with the Functional Activities Questionnaire (FAQ). The FAQ includes 10 items which are scored on a scale from 0 to 3 where 0 = normal and 3 = dependent. Total scores range from 0 to 30 and lower scores indicate that the respondent is able to perform daily activities. A score of 9 (where the person is dependent in 3 activities) is used as a cut-point indicating impairments with functioning.
Time Frame: Day 180
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Protocol | Control Protocol
Number analyzed (Participants) | 252 | 249
score on a scale | 9.5 (10.8) | 7.7 (9.2)

17. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Depression 6
Description: Depression is assessed with the PROMIS Depression 6 instrument. This tool includes 6 items with response options on a scale of 1 to 5. Total raw scores range from 6 to 30 with higher scores indicating greater symptoms of depression.
Time Frame: Day 180
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Protocol | Control Protocol
Number analyzed (Participants) | 252 | 249
score on a scale | 11.9 (6.3) | 11.9 (5.9)

18. Secondary Outcome: Posttraumatic Stress Disorder-8 (PTSD-8) Score
Description: Posttraumatic Stress Disorder (PTSD) is assessed with the Posttraumatic Stress Disorder - 8 instrument. The PTSD-8 includes 8 items which are answered on a 4 point scale where 01 = not at all and 3 = all of the time. Total scores range from 0 to 24 where higher scores indicate greater symptoms of PTSD.
Time Frame: Day 180
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Protocol | Control Protocol
Number analyzed (Participants) | 252 | 249
score on a scale | 5.7 (5.8) | 5.2 (5.1)

19. Secondary Outcome: EuroQol, 5 Dimension (EQ-5D) Visual Analog Scale Score
Description: Quality of life is assessed with the Visual Analog Scale of the EuroQol, 5 dimension (EQ-5D) questionnaire. The EQ-5D asks about 5 dimensions of health (mobility, self-care, usual activities, pain, and depression). The questionnaire includes a visual analog scale where respondents rate their current health where 0 = worst health imaginable and 100 = best health imaginable.
Time Frame: Day 180
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Protocol | Control Protocol
Number analyzed (Participants) | 252 | 249
units on a scale | 66 (22) | 67 (22)

ADVERSE EVENTS:
Time Frame: Adverse events potentially associated with the study treatment and serious adverse events were monitored from the time of randomization up to Day 30. Mortality was recorded from the time of randomization up to Day 180.
Description: Adverse events that were not considered serious or potentially associated with the treatment were not recorded.
Arm/Group | Treatment Protocol | Control Protocol
All-Cause Mortality (participants affected / at risk) | 102/252 | 94/249
Serious Adverse Events (participants affected / at risk) | 0/252 | 0/249
Other Adverse Events (participants affected / at risk) | 2/252 | 0/249
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Protocol (N=252) | Control Protocol (N=249)
Hemorrhagic shock due to hemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Worsening of renal function (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-22): https://cdn.clinicaltrials.gov/large-docs/50/NCT03509350/Prot_SAP_000.pdf